CLINICAL TRIAL: NCT03218982
Title: A Culturally-Relevant Approach to Reducing Dementia Caregiver Stress in an Underserved Population
Brief Title: Vietnamese Caregiver Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 823071; K01AG052646 (NIH)
Record Dates: First submitted 2017-06-12; First posted 2017-07-17 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Alzheimer's Disease (Incl Subtypes); Cognitive Impairment
Keywords: Caregiver; Vietnamese; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Families will then be randomized (as a team) to either the active intervention or the control condition. Caregivers in the active intervention will then be scheduled for six weekly intervention sessions, lasting about 2 hours each. Following the completion of the sessions, primary caregivers will complete assessment measures (that they completed at baseline) immediately after the intervention (post) and at three months. This is expected to take one hour for each assessment. Primary caregivers assigned to the control condition will also complete these assessment measures around the same those in the active intervention complete them. These caregivers will also have the option of participating in the active intervention after the three-month follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention (Experimental): Six weekly intervention sessions (2 hours, each) that include enhanced psycho-education and discussion of AD and cultural impacts on beliefs about dementia and caregiving, management of problem behaviors, facilitation of support seeking, and mindful Tai Chi.
  Interventions: Behavioral: Enhanced psycho-education about dementia and caregiving
- Control (No Intervention): Participants will receive educational materials/pamphlets on dementia and occasional phone-calls by research assistants to maintain contact, as is the standard of care in most caregiver intervention studies.

INTERVENTIONS:
Behavioral: Enhanced psycho-education about dementia and caregiving — Enhanced psycho-education re dementia and caregiving helping family members come to shared understanding of the nature and cause of dementia. Discussion of cultural values in Vietnamese and American cultures and how this can influence perceptions of dementia and caregiving strategies will help family members who disagree on the etiology of dementia and strategies for care to empathize with each other's perspective. Other sessions will teach skills to develop self-efficacy in dealing with patient symptoms, to access resources (e.g., in-home support), and to gain family support in culturally-congruent ways. Mindful Tai Chi is rooted in East Asian traditions and philosophies that promote balance and healing of the mind and body, thus addressing holistic beliefs Vietnamese have about wellness.
  Other Names: management of problem behaviors; facilitation of support-seeking; mindful Tai Chi
  Arms: Active Intervention

SUMMARY:
The purpose of this study is to develop and implement a culturally-appropriate intervention to reduce stress in Vietnamese dementia caregivers. A pilot intervention will be done to test the feasibility and acceptability of the intervention in a community setting. This will be done by randomly assigning a family triad (primary caregiver, secondary caregiver, and their care recipient) into an active intervention or a control condition and monitoring findings at baseline, post-intervention, and at three months.The intervention will consist of multiple components -enhanced psycho-education that includes discussion of Alzheimer's Disease (AD) and cultural impacts on beliefs about dementia and caregiving, management of problem behaviors, facilitation of support seeking, and mindful Tai Chi. A secondary caregiver who the primary caregiver identifies as providing him/her with the most support will be invited to join all components, but the intervention will be flexible depending on caregivers' needs/preferences. The care recipient is not required to join the sessions but will be able to if he/she or the family wishes. During the intervention, community partners will provide respite care for the care recipient.

DETAILED DESCRIPTION:
Twenty-four (24) caregivers, the identified secondary caregiver, and a care recipient will be randomly assigned into the active intervention or a control condition: 16 triads in the intervention condition, 8 in the control.

For the primary caregivers: Primary caregivers will attend six weekly intervention sessions lasting 2 hours each. Based on previous Randomized Controlled Trials (RCTs) of a successful behavior change (i.e., smoking cessation) intervention in Vietnamese using only 2-3 sessions, six sessions were chosen as a middle ground. In the first 45 minutes, primary caregivers and a secondary caregiver (who the primary caregiver identifies) will participate in family psycho-education delivered by a Master's level trained, bilingual facilitator. Each group will consist of no more than four dyads (4 different groups totaling 16 dyads). The curriculum will be adapted based on what the Alzheimer's Association and REACH II have successfully used as well as what the University of California (UC) Davis Alzheimer's Disease Center (ADC) has implemented. The sessions will cover the following: a clinical model of dementia and helping family members come to a shared understanding of the nature and cause of dementia. The innovative component is a discussion of cultural values typical of individuals in Vietnamese and American cultures and how this can influence perceptions of dementia and caregiving strategies. This is important because it will help family members who disagree on the etiology of dementia and strategies for care to empathize with each other's perspective. Subsequent sessions will help caregivers learn skills and develop self-efficacy in dealing with patient symptoms, accessing resources (e.g., in-home support), and gaining family support in culturally-congruent ways. Facilitating the use of formal and informal support is a critical piece as Vietnamese caregivers may be looking for basic and concrete assistance rather than help in coping with caregiving.

The last part of the intervention is mindful Tai Chi that was chosen for several reasons. In a recent review and meta-analysis, Tai Chi showed beneficial effects on depression, anxiety, stress management, and self-efficacy. Second, Tai Chi is rooted in East Asian traditions and philosophies that promote balance and healing of the mind and body, thus addressing holistic beliefs Vietnamese have about wellness. An RCT of Tai Chi recently was successfully completed in Vietnam, demonstrating its growing acceptance in the Vietnamese population. The protocol will be adapted to meet caregivers' needs and highlight meditation that involves accepting stressful circumstances, thus capitalizing on emotion regulation strategies.

For the care recipients: Care recipients will receive the Montreal Cognitive Assessment (MoCA) measure to assess their mental status at baseline. The purpose of the Quality of Life - Alzheimer's Disease (QoL-AD) measure is to assess the caregiver intervention affects the care recipient's quality of life. The total time to complete these questionnaires is about 30 minutes per session.

Participants not randomized to the active intervention will receive educational materials/pamphlets on dementia and occasional phone-calls by research assistants to maintain contact, as is the standard of care in most caregiver intervention studies. Including a control condition will allow for mirroring of the actual larger trial as closely as possible, and also ascertain the feasibility of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers will be included if they (a) are Vietnamese; (b) are age 21+; (c) speak Vietnamese and/or English (d) provide day-to-day, hands on care to a family member with Alzheimer's disease (AD) or cognitive impairment related to AD (e) have at least one family member who will also participate in the intervention; (f) volunteer informed consent; (g) are physically able to participate; and (g) expect to stay in the Sacramento area for the duration of the study
* Care recipients will be included if they are (a) Vietnamese; (b) are age 21+; (c) have reported Alzheimer's disease (AD) or cognitive impairment related to AD; (d) have at least one caregiver who is participating in the intervention (e) volunteer informed consent or surrogate consent, and (f) expect to stay in the Sacramento area for the duration of the study

Exclusion Criteria:

* If the care recipient expresses dissent to participation or to the use of surrogate consent, then he/she will be excluded from the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Randomization | assessed once all 3-month follow-ups are complete
  % of eligible dyads who agree to randomization
Retention | assessed once all 3-month follow-ups are complete
  Retention in both arms of the study; Note: no formal assessment tool will be used - this will be assessed via number of participants retained
Caregiver Intervention Adherence | assessed at end of study, once all 3-month follow-ups are complete
  % of dyads engaging in the initial session, % completing at least 3 sessions, and % completing all sessions
Treatment Fidelity | assessed once all 3-month follow-ups are complete
  Extent to which the facilitator adheres to the intervention protocol, as measured by a self-report checklist, with a goal of 85% adherence to key elements
Administration of Study Measures | assessed at end of study, once all 3-month follow-ups are complete
  % of baseline, post-, and 3-month assessments completed (considering length of assessments and completeness of collected data
Acceptability | 2 years
  Assessed through a questionnaire and interview assessing the perceptions of the intervention by primary and secondary caregivers, CBO staff/administrators, and interventionists.

SECONDARY OUTCOMES:
Alzheimer's Disease Knowledge Scale (ADKS) | Baseline, 6-weeks (Post-intervention), 3 months post-intervention
  This scale assesses knowledge about AD. The scale has 30 statements. Subjects are asked to rate each statement as True or False.
Caregiver Self-Efficacy | Baseline, 6-weeks (Post-intervention), 3 months post-intervention
  Asks the caregiver about how confident in their ability to keep up their own activities and also respond to caregiving situations. The Scale includes 10 items, and asks caregivers to rate their confidence in handling situations on a scale from 1 to 10.
Center for Epidemiological Studies Depression (CES-D) scale | Baseline, 6-weeks (Post-intervention), 3 months post-intervention
  This is a self-report depression scale that asks how many times during the past week a person has felt symptoms of depression. There are 20 items.
Zarit Burden Inventory (ZBI) | Baseline, 6-weeks (Post-intervention), 3 months post-intervention
  This is a caregiver self-report measure that contains 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always).
Quality of Life - Alzheimer's Disease (QoL-AD) | Baseline, 6-weeks (Post-intervention), 3 months post-intervention
  The QOL-AD is a brief, 13-item measure designed specifically to obtain a rating of the patient's Quality of Life from both the patient and the caregiver. It was developed for individuals with dementia, based on patient, caregiver, and expert input, to maximize construct validity, and to ensure that the measure focuses on quality of life domains thought to be important in cognitively impaired older adults. It uses simple and straightforward language and responses & includes assessments of the individual's relationships with friends and family, concerns about finances, physical condition, mood, and an overall assessment of life quality.
Perceived Stress Scale | Baseline, 6-weeks (Post-intervention), 3 months post-intervention
  This scale asks subjects about how often they have felt or thought about 10 items during the past month.

CONTACTS AND LOCATIONS:
Overall Officials: Oanh Meyer, PhD, MAS, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Meyer OL, Nguyen KH, Dao TN, Vu P, Arean P, Hinton L. The Sociocultural Context of Caregiving Experiences for Vietnamese Dementia Family Caregivers. Asian Am J Psychol. 2015 Sep;6(3):263-272. doi: 10.1037/aap0000024. Epub 2015 Jun 15. PMID 26617956
- [Background] Resnick B, Ory MG, Hora K, Rogers ME, Page P, Bolin JN, Lyle RM, Sipe C, Chodzko-Zajko W, Bazzarre TL. A proposal for a new screening paradigm and tool called Exercise Assessment and Screening for You (EASY). J Aging Phys Act. 2008 Apr;16(2):215-33. doi: 10.1123/japa.16.2.215. PMID 18483443
- [Background] Callahan CM, Unverzagt FW, Hui SL, Perkins AJ, Hendrie HC. Six-item screener to identify cognitive impairment among potential subjects for clinical research. Med Care. 2002 Sep;40(9):771-81. doi: 10.1097/00005650-200209000-00007. PMID 12218768
- [Background] Jorm AF, Jacomb PA. The Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE): socio-demographic correlates, reliability, validity and some norms. Psychol Med. 1989 Nov;19(4):1015-22. doi: 10.1017/s0033291700005742. PMID 2594878
- [Background] Carpenter BD, Balsis S, Otilingam PG, Hanson PK, Gatz M. The Alzheimer's Disease Knowledge Scale: development and psychometric properties. Gerontologist. 2009 Apr;49(2):236-47. doi: 10.1093/geront/gnp023. Epub 2009 Mar 25. PMID 19363018
- [Background] Fortinsky RH, Kercher K, Burant CJ. Measurement and correlates of family caregiver self-efficacy for managing dementia. Aging Ment Health. 2002 May;6(2):153-60. doi: 10.1080/13607860220126763. PMID 12028884
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] Schulz R, Burgio L, Burns R, Eisdorfer C, Gallagher-Thompson D, Gitlin LN, Mahoney DF. Resources for Enhancing Alzheimer's Caregiver Health (REACH): overview, site-specific outcomes, and future directions. Gerontologist. 2003 Aug;43(4):514-20. doi: 10.1093/geront/43.4.514. No abstract available. PMID 12937330
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Phan T, Steel Z, Silove D. An ethnographically derived measure of anxiety, depression and somatization: the Phan Vietnamese Psychiatric Scale. Transcult Psychiatry. 2004 Jun;41(2):200-32. doi: 10.1177/1363461504043565. PMID 15446721